CLINICAL TRIAL: NCT00280696
Title: A Double-blind, Randomized, Placebo-controlled 5 Parallel Groups, Confirmatory Trial on the Efficacy and Safety of Levetiracetam Used as add-on Therapy at Doses of 0.5 to 3 g/Day in Patients From 16 to 65 Years With Epilepsy With Partial Onset Seizures Under Treatment With 1 to 3 Anti-epileptic Drug(s)
Brief Title: A Double-blind Confirmatory Trial of Levetiracetam in Epilepsy Patients With Partial Onset Seizures
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Japan Co. Ltd. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: N01221; 2014-004333-57 (EudraCT Number)
Record Dates: First submitted 2006-01-19; First posted 2006-01-23 (Estimated); Last update posted 2015-02-11 (Estimated); Status verified 2015-02

CONDITIONS: Epilepsies, Partial
Keywords: Epilepsies, Partial,; Keppra, levetiracetam
MeSH Terms: conditions — Epilepsies, Partial | interventions — Levetiracetam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Lev 0.5 g (Experimental): Levetiracetam 0.5 g/day as add-on therapy to ongoing treatment with 1 to 3 AED(s) administered orally twice daily (in the morning and evening).
  Interventions: Drug: Levetiracetam 250 mg
- Lev 1 g (Experimental): Levetiracetam 1 g/day as add-on therapy to ongoing treatment with 1 to 3 AED(s) administered orally twice daily (in the morning and evening).
  Interventions: Drug: Levetiracetam 250 mg; Drug: Levetiracetam 500 mg
- Lev 2 g (Experimental): Levetiracetam 2 g/day as add-on therapy to ongoing treatment with 1 to 3 AED(s) administered orally twice daily (in the morning and evening).
  Interventions: Drug: Levetiracetam 250 mg; Drug: Levetiracetam 500 mg
- Lev 3 g (Experimental): Levetiracetam 3 g/day as add-on therapy to ongoing treatment with 1 to 3 AED(s) administered orally twice daily (in the morning and evening).
  Interventions: Drug: Levetiracetam 250 mg; Drug: Levetiracetam 500 mg
- Placebo (Placebo Comparator): Placebo tablets as add-on therapy to ongoing treatment with 1 to 3 AED(s) administered orally twice daily (in the morning and evening).
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Levetiracetam 250 mg — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 250 mg
  * Route of Administration: Oral Use
  Other Names: Keppra
  Arms: Lev 0.5 g; Lev 1 g; Lev 2 g; Lev 3 g
Drug: Levetiracetam 500 mg — * Active Substance: Levetiracetam
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 500 mg
  * Route of Administration: Oral Use
  Other Names: Keppra
  Arms: Lev 1 g; Lev 2 g; Lev 3 g
Other: Placebo — * Active Substance: Placebo
  * Pharmaceutical Form: Film-coated tablet
  * Concentration: 250 mg and 500 mg
  * Route of Administration: Oral Use
  Arms: Placebo

SUMMARY:
A double-blind, randomized, multicenter, placebo controlled 5 parallel groups, confirmatory trial to evaluated the efficacy and safety of levetiracetam used as adjunctive treatment in patients from 16 to 65 years with epilepsy suffering from partial onset seizures.

ELIGIBILITY:
Inclusion Criteria:

Epileptic patients who fulfill the following criteria are eligible for inclusion in the study:

* Subjects aged from 16 to 65 years at the acquisition of informed consent to the trial participation
* Seizure type: subjects with epileptic seizures which were diagnosed as partial seizures more than 2 years ago according to "Clinical and electroencephalographic classification of epileptic seizures (1981)" defined by the International League Against Epilepsy (ILAE) and confirmed with an EEG that has been performed within 1 year before Screening or at the Screening Visit
* Subjects whose previous therapy before screening involved at least two standard anti-epileptic drugs (AEDs) for partial seizures, and in whom it can be confirmed that the doses met the daily dose specified for the treatment of epilepsy in the package insert and that the therapy has been continued for at least 3 months
* Frequency of epileptic seizures: subjects experiencing partial seizures at least 12 times in 12 weeks during the Baseline Period (Week -12 to Week 0) and at least twice in every 4 weeks

Exclusion Criteria:

The following patients are not eligible for inclusion into the study:

* Subjects who were diagnosed with status epilepticus within 3 months before screening
* Subjects with no partial seizures of which frequency was measured during the Baseline Period
* Subjects who underwent surgery for epilepsy within 2 years before Screening or who were scheduled to undergo brain surgery during the study period and within 4 weeks after the completion of this study
* Subjects with a history of oral treatment with Levetiracetam (LEV)

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2005-11; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Percent reduction from Baseline in partial (Type I) seizure frequency per week over the Evaluation Period | From Baseline to the 12-week Evaluation Period

SECONDARY OUTCOMES:
Partial (Type I) seizure frequency per week over the Evaluation Period | 12-week Evaluation Period
Partial (Type I) seizure responder rates (50 %, 75 %) over the Evaluation Period | From Baseline to the 12-week Evaluation Period
Seizure freedom over the Evaluation Period | 12-week Evaluation Period
Categorized percentage reduction from Baseline in partial (Type I) seizure frequency per week over the Evaluation Period | From Baseline to the 12-week Evaluation Period
Percentage reduction from Baseline in seizure frequency per week by seizure subtype (IA, IB, IC, IA + IB, other) over the Evaluation Period | From Baseline to the 12-week Evaluation Period

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (37):
- Japan (37):
  - Aichi-gun, Aichi-ken
  - Nagoya, Aichi-ken
  - Nayoga, Aichi-ken
  - Hirosaki, Aomori
  - Chiba, Chiba
  - Fukuoka, Fukuoka
  - Kitakyushu, Fukuoka
  - Kurume, Fukuoka
  - Gifu, Gihu
  - Fukuyama, Hiroshima
  - Hiroshima, Hiroshima
  - Asahikawa, Hokkaido
  - Hakodate, Hokkaido
  - Sapporo, Hokkaido
  - Kobe, Hyōgo
  - Kahoku-gun, Ishikawa-ken
  - Kagoshima, Kagoshima-ken
  - Kikuchi-gun, Kumamoto
  - Kyoto, Kyoto
  - Sendai, Miyagi
  - Miyazaki, Miyazaki
  - Nagaoka, Nagaoka
  - Ōmura, Nagasaki
  - Niigata, Niigata
  - Okayama, Okayama-ken
  - Izumi, Osaka
  - Neyagawa, Osaka
  - Osaka, Osaka
  - Suita, Osaka
  - Shizuoka, Shizuoka
  - Kawachi-gun, Tochigi
  - Kodaira, Tokyo
  - Tokyo, Tokyo
  - Toyama, Toyama
  - Yamagata, Yamagata
  - Ube, Yamaguchi
  - Kobe

REFERENCES:
- [Derived] Inoue Y, Yagi K, Ikeda A, Sasagawa M, Ishida S, Suzuki A, Yoshida K; Japan Levetiracetam N01221 Study Group. Efficacy and tolerability of levetiracetam as adjunctive therapy in Japanese patients with uncontrolled partial-onset seizures. Psychiatry Clin Neurosci. 2015 Oct;69(10):640-8. doi: 10.1111/pcn.12300. Epub 2015 May 13. PMID 25854635